CLINICAL TRIAL: NCT00953264
Title: Hormonal and Metabolic Effects of Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Professor Joachim Spranger, Professor, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EA4/042/07
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2016-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- life style intervention (Experimental)
  Interventions: Behavioral: lifestyle

INTERVENTIONS:
Behavioral: lifestyle — lifestyle intervention, including diet, physical activity and behavioral changes

SUMMARY:
The investigators here propose to evaluate the hormonal and metabolic effects of weight loss, including evaluation of changes in several tissues.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 27 kg/m2 (adults)

Exclusion Criteria:

* pregnancy, breastfeeding
* patients with:

  * heart failure
  * impaired hepatic or renal function
  * anaemia
  * disturbed coagulation
  * infection, malabsorption
  * severe hypertension
  * any other endocrine disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2007-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
hormonal and metabolic changes during weight loss | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Charite, Berlin, Germany